CLINICAL TRIAL: NCT00974181
Title: The European Cobalt STent With Antiproliferative for Restenosis Trial (EuroSTAR Trial)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Collaborators: Conor Medsystems (Industry)
Responsible Party: Sidney A. Cohen, MD, PhD/Vice President, Medical Affairs, Cordis Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EUS08; EUROSTAR
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2010-05-17 (Estimated); Status verified 2010-05

CONDITIONS: Treatment of Symptomatic Ischemic Heart Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conor Medsystems COSTAR™ stent (10 µg Paclitaxel) (Active Comparator): Conor Medsystems COSTAR™ stent loaded with the antiproliferative compound paclitaxel (10 µg), pre-mounted on a rapid exchange, percutaneous transluminal coronary angioplasty balloon catheter.
  Interventions: Device: Conor Medsystems COSTAR™ stent (10 µg Paclitaxel)
- Conor Medsystems COSTAR™ stent (30 µg Paclitaxel) (Active Comparator): Conor Medsystems COSTAR™ stent loaded with the antiproliferative compound paclitaxel (30 µg), pre-mounted on a rapid exchange, percutaneous transluminal coronary angioplasty balloon catheter.
  Interventions: Device: Conor Medsystems COSTAR™ stent (30 µg Paclitaxel)

INTERVENTIONS:
Device: Conor Medsystems COSTAR™ stent (10 µg Paclitaxel) — Intervention will consist of percutaneous coronary intervention for treatment of one or more de-novo coronary lesion(s) using standard coronary intervention techniques. Intervention in this arm will include treatment with the CoStar™ Paclitaxel-Eluting Coronary Stent System (10 µg Paclitaxel)
  Arms: Conor Medsystems COSTAR™ stent (10 µg Paclitaxel)
Device: Conor Medsystems COSTAR™ stent (30 µg Paclitaxel) — Intervention will consist of percutaneous coronary intervention for treatment of one or more de-novo coronary lesion(s) using standard coronary intervention techniques. Intervention in this arm will include treatment with the CoStar™ Paclitaxel-Eluting Coronary Stent System (30 µg Paclitaxel)
  Arms: Conor Medsystems COSTAR™ stent (30 µg Paclitaxel)

SUMMARY:
Two consecutive cohorts of subjects were each treated with the CoStar stent loaded with a different paclitaxel dose regimen. The first 145 subjects (Arm I), enrolled between 20 January 2004 and 26 May 2004, were treated with 10 µg paclitaxel and the subsequent 137 subjects (Arm II), enrolled between 15 December 2004 and 9 March 2005, were treated with 30 µg paclitaxel. Both dose formulations eluted over 30 days (in-vitro).

Subjects in both arms completed clinical follow-up at 1, 6 and 12 months post-index procedure, with angiographic follow-up at 6 months as outlined in the original study protocol.

Based on results from previous studies and the initial EuroSTAR Trial results, Conor Medsystems decided to pursue the dosage used in Arm I, 10 μg/30 days, as the commercial dose formulation for the CoStar® stent. The EuroSTAR Trial addendum was proposed for the purpose of evaluating the long-term clinical outcomes of the CoStar stent.

DETAILED DESCRIPTION:
The EuroSTAR Trial (European Cobalt STent with Antiproliferative for Restenosis Trial) is a prospective, multi-center, two-arm study to evaluate the safety and performance of the CoStar® stent for the treatment of symptomatic ischemic heart disease attributable to stenotic de novo lesions of the native coronary arteries that are amenable to treatment by percutaneous stenting.

ELIGIBILITY:
Inclusion Criteria:

All subjects admitted for PCI should be screened for study eligibility.

The subject must meet the following criteria for inclusion into the Study:

1. Subject is ≥ 18-80 years of age,
2. Subject understands the risks, benefits and alternatives to Percutaneous Coronary Intervention (PCI) and has signed the Informed Consent as approved by the Institution for the implantation of the COSTAR™ stent,
3. Subject is willing and able to return for the clinical and angiographic follow up,
4. Subject is an acceptable candidate for planned PCI,
5. Subject has stable or unstable angina pectoris (CCS Classification I or greater), or a positive functional study for ischemia,
6. Subject is male, or female subject is post-menopausal or of non-child bearing potential, and/or has a negative pregnancy test at the time of PCI, and
7. No other treatments are planned within 30 days of the procedure.

   Up to two lesions may be treated using the COSTAR™ stent per study subject, either two discreet lesions in one vessel separated by > 20mm or two discreet lesions in two native coronary arteries. Upon coronary angiography at the time of PCI, each lesion under consideration for treatment must meet the following angiographic criteria for inclusion into the study:
8. The target lesion is a de-novo lesion in a native coronary artery that has not been treated with any previous interventional procedure,
9. The target lesion meets the following angiographic criteria by visual assessment of the Investigator:

   1. The target lesion stenosis must be between 50-99%,
   2. The target reference vessel diameter is between 2.5 mm and 3.5mm,
   3. The lesion length is ≤25 mm, and
   4. Target vessel Thrombolysis in Myocardial Infarction (TIMI) flow must be grade 1 or higher.

Exclusion Criteria:

1. Subject has a left ventricular ejection fraction of <30%,
2. Subject has an imminent co-morbid illness (i.e., life expectancy less than 2 years),
3. Subject has experienced an acute myocardial infarction (MI) 72 hours prior to the procedure, as defined either by the presence of a new Q wave in 2 or more contiguous leads, or by a CK greater than two times site upper limit normal value with presence of CKMB greater than the site upper limit normal value,
4. Subject has a known allergy or hypersensitivity to cobalt steel, contrast medium, heparin, or aspirin,
5. Subject has a history of an allergic reaction of hypersensitivity to paclitaxel or drugs in a similar class,
6. Subject is contraindicated for or unwilling to take aspirin and clopidogrel or ticlopidine,
7. Subject has known peptic ulcer with recent (<3 months GI bleeding,
8. Subject has had a cerebrovascular event (CVA) or transient ischemic attack (TIA) within the prior 6 months,
9. Subject has renal failure defined as a serum creatinine level >2.5 mg/dL,
10. Subject is in cardiogenic shock,
11. Subject has unstable ventricular arrhythmia,
12. Subject is currently enrolled in another investigational drug or device trial,
13. Subject has undergone PCI or CABG surgery within 30 days of the procedure, and
14. Subject is unable to comply with the follow up requirements, or would be unreliable for follow up documentation.

    Upon coronary angiography at the time of PCI, the lesion was excluded from the study if any of the following angiographic criteria were met:
15. More than 2 lesions required treatment at the time of the procedure
16. Presence of intraluminal thrombus in the target vessel
17. The target lesion involved a bifurcation where the adjacent vessel was greater than 2 mm in diameter requiring intervention
18. Patient had an evolving myocardial infarction as evidenced by persistent new ECG changes during PCI (defined as new ST segment elevation or depression of > 1.0 mm for > 30 min).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2004-01; Primary Completion 2005-05 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint Angiographic late loss at 6 months as measured by Quantitative Coronary Analysis (QCA) | 6 months post-procedure

SECONDARY OUTCOMES:
Endpoints are binary angiographic restenosis and vessel diameter stenosis measured by QCA | 30 days, 6 months, and 12 months post-procedure
Clinical endpoints include device, lesion, and procedural success rates associated with implantation procedure | 30 days, 6 months, and 12 months post-procedure
Safety endpoint consists of composite of major adverse cardiac events | 30 days, 6 months, 1, 2, 3, 4 and 5 year post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Colombo, MD, Principal Investigator — EMO Centro Cuore Columbus
Locations (1):
- EMO Centro Cuore Columbus, Milan, Italy